CLINICAL TRIAL: NCT04599504
Title: Pharmacological and Behavioral Treatments to Treat Loss-of-Control Eating and Improve Weight Outcomes After Bariatric Surgery: Medication Change for Non-Responders (Stage 2b)
Brief Title: Pharmacological and Behavioral Treatment After Bariatric Surgery: Medication Change for Non-Responders (Stage 2b)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000029057b; 5R01DK126637-02 (NIH)
Record Dates: First submitted 2020-10-21; First posted 2020-10-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Loss-of-control Eating; Obesity/Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Lisdexamfetamine Dimesylate; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lisdexamfetamine dimesylate (Experimental)
  Interventions: Drug: Lisdexamfetamine Dimesylate (Medication)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate (Medication) — Medication will be taken daily in pill form.
  Other Names: Vyvanse
  Arms: Lisdexamfetamine dimesylate
Other: Placebo — Placebo will be inactive and taken daily in pill form.
  Arms: Placebo

SUMMARY:
This study will test the effectiveness of lisdexamfetamine medication as a treatment for loss-of-control eating and weight following bariatric surgery. This is a controlled test of whether, amongst non-responders to acute treatments, lisdexamfetamine medication results in superior outcomes compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Be in the age range ≥18 years of age and <65 years of age.
* Have had laparoscopic Roux-en-Y gastric bypass or sleeve gastrectomy
* Approximately ten months post-surgery
* Experienced regular loss of control eating about six months after bariatric surgery, and were considered treatment non-responders to a four-month treatment trial of medication and/or BWL
* Be an otherwise healthy subject without uncontrolled medical problems, as determined by the study physician and medical co-investigators (physical examination, laboratory studies).
* Read, comprehend, and write English at a sufficient level to complete study-related materials.
* Provide a signed and dated written informed consent prior to study participation.
* Be available for participation in the study for up to 15 months (3-month treatment plus 12-month follow up).

Exclusion Criteria:

* Has a predisposition to seizures (e.g., subject with a history or evidence of seizure disorder, febrile seizures during childhood, brain tumor, cerebrovascular disease, or significant head trauma; has a family history of idiopathic seizure disorder or is currently being treated with medications or treatment regimens that lower seizure threshold).
* Has a history of anorexia nervosa or history of bulimia nervosa.
* Is currently using other medications for weight loss.
* Has a co-existing psychiatric condition that requires hospitalization or more intensive treatment (such as bipolar mood disorders, psychotic illnesses, or severe depression)
* Has untreated hypertension with a seated systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg, or heart rate > 100 beats/minute.
* Has a history of congenital heart disease, cardiovascular disease, cardiac arrhythmias requiring medication, or a history of cerebrovascular pathology including stroke.
* Has current uncontrolled hypertension.
* Has current uncontrolled Type I or Type II diabetes mellitus.
* Has untreated hypothyroidism with a TSH > 1.5 times the upper limit of normal for the test laboratory with repeat value that also exceeds this limit.
* Has gallbladder disease.
* Has a history of severe renal, hepatic, neurological, chronic pulmonary disease, or any other unstable medical disorder.
* Is currently in active treatment for eating or weight loss.
* Is currently participating in another clinical study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.
* Is breast-feeding or is pregnant or is not using a reliable form of birth control.
* Reports active suicidal or homicidal ideation.
* Previous history of problems with LDX or other stimulants.
* Has a history of allergy or sensitivity to LDX or other stimulant medications.
* Current medication contraindicated with study medication.
* Any current psychostimulant use or any medication for ADHD.
* History or current alcohol or substance use disorder (smoking will not be exclusionary)
* Is currently taking MAOI medication, SSRI medication, or strong inhibitors of CYP2D6

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Loss-of-Control Eating Frequency | From baseline interview at study enrollment to after the 12-week treatment
  Loss-of-control eating frequency is a continuous variable of loss-of-control eating episodes assessed using the Eating Disorder Examination interview; Loss-of-control eating frequency will be based on the past 28 days and defined as loss-of-control eating episodes per month.
Loss-of-Control Eating Frequency | From post-treatment to the 6-month follow-up
  Loss-of-control eating frequency is a continuous variable of loss-of-control eating episodes assessed using the Eating Disorder Examination interview; Loss-of-control eating frequency will be based on the past 28 days and defined as loss-of-control eating episodes per month.
Loss-of-Control Eating Frequency | From post-treatment to the 12-month follow-up
  Loss-of-control eating frequency is a continuous variable of loss-of-control eating episodes assessed using the Eating Disorder Examination interview; Loss-of-control eating frequency will be based on the past 28 days and defined as loss-of-control eating episodes per month.
Body Mass Index (BMI) | From baseline at study enrollment to after the 12-week treatment
  BMI is calculated using measured height and weight
Body Mass Index (BMI) | From post-treatment to the 6-month follow-up
  BMI is calculated using measured height and weight
Body Mass Index (BMI) | From post-treatment to the 12-month follow-up
  BMI is calculated using measured height and weight

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Grilo, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No